CLINICAL TRIAL: NCT05131906
Title: Assessing the Use of Lasers on Shoes for Freezing of Gait in People With Parkinson's Disease: A Pilot Study
Brief Title: Laser Shoes for Freezing in People With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northern Arizona University (Other)
Collaborators: FY2020 Research Bridge (Unknown); Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1550436-1
Record Dates: First submitted 2021-05-20; First posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Parkinson Disease
Keywords: Freezing of gait; laser shoes; Parkinson's disease; External cueing; Parkinsonian Disorder; Movement Disorders; Neurodegenerative Diseases; Freezing
MeSH Terms: conditions — Parkinson Disease; Movement Disorders; Neurodegenerative Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- People with Parkinson's disease on medication who freeze (Experimental): We will be testing each of the 15 participants both with and without the removeable lasers on their shoes.
  Interventions: Device: gait task and activity of daily living task

INTERVENTIONS:
Device: gait task and activity of daily living task — use of lasers on shoes to potentially minimize freezing of gait
  Other Names: A gait task and activity of daily living task without laser shoe attachment

SUMMARY:
The purpose of this study is to assess the effectiveness of the visual cues of a wearable device in preventing freezing of gait (FOG) in those with PD.The aim is to investigate the impact of laser shoe attachments on gait in single and dual-tasking scenarios, as well as "real-world" mobility scenarios, in people with PD who freeze. For this study, participants will wear sensors on their feet, hips, chest, and head to show stride length, foot angle, and foot height, and head position during different gait assessments. The patients will do the gait assessments without the laser shoes and with the laser shoes to determine how the laser shoes affect freezing of gait. The gait assessments include having the patient complete a two minute walk, two minute walk with another task (reciting every other letter of the alphabet), obstacle course, obstacle course with another task (reciting every other letter of the alphabet), and quickly turning in place. The assessments are activities that are performed in everyday activities so there are no risks associated with these requested tasks. These activities will be done in a lab at the Phoenix Biomedical Campus. Safety for the participants will be monitored by placing a belt around the waist of the participant with a member of the research personnel close by in case the participant demonstrated a shift in their balance. The research member can use the belt to provide stability and secure the participant, preventing them from further loss of balance. Moreover, three different activities of daily living (ADL's) will be assessed with and without the laser shoes in a simulated apartment environment located at the Phoenix Biomedical campus. The ADL's include walking from the bed to the kitchen, walking from the living room to the kitchen and making tea in the microwave, and answering the door. The activities to be done in the apartment setting will be video-recorded and analyzed. Some participants will be given the laser shoes to take home and use for one week. The same protocol explained above will be used to assess freezing of gait after this one week in those selected participants. To assess retention of improvements, the participants who took the laser shoes home will also be given the same protocol two days later (after not having used the laser shoes during that time). Participants will also complete surveys for quality of life, freezing and gait and cognitive function. A standard test for balance will also be conducted.

DETAILED DESCRIPTION:
15 individuals with Parkinson's Disease will complete two tasks: a gait task and an activity of daily living (ADL) task both with and without the use of laser shoe attachment. The gait task involves 5 separate scenarios: 2 min walk with a single and dual-task trial, obstacle course with a single and dual-task trial, and a quick turn-in-place. For the dual-task trials, participants will complete the 2 min walk and obstacle course scenarios in addition to a cognitive task (e.g. reciting the alphabet every other letter). During the single-task trials for the 2 min walk and obstacle course, participants will complete these activities without a cognitive task. Participants will also be required to fill out surveys for quality of life, balance and freezing of gait. A standard test for balance will be conducted (MiniBEST). Participants will be assessed using the UPDRS in order to categorize the level of Parkinson's Disease. Permission and training for use of the UPDRS will be obtained prior to testing participants.

The ADL task involves three "real-world" mobility scenarios, in which participants will be asked to: walk from the bedroom to the bathroom and also the kitchen, make tea in the kitchen, and move from the couch to answer the front door.

For both tasks, gait will be characterized during each scenario using inertial sensors (OPALs). Outcomes will include step length, foot angle and foot height (clearance from floor) and head movement. To characterize functional movements we will video movements during all scenarios for both tasks. Outcomes will be the number and temporal length of each freezing event, to be determined by a movement disorders neurologist.

A subset of participants (n=3) will use the sensors at home for 1 week, and return to the lab for gait and functional task assessment. They will return after a 2-day washout (no sensors) to assess retention of improvements from the 1-week exposure.

ELIGIBILITY:
Inclusion Criteria:

* People with PD who exhibit freezing, on medications

Exclusion Criteria:

* People who are non-ambulatory

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-12-12 (Actual); Primary Completion 2022-07-14 (Estimated); Study Completion 2022-07-14 (Estimated)

PRIMARY OUTCOMES:
Freezing Severity | 4 hours
  The severity of freezing during a gait task, as quantified by review of a video of the movement, assessed by a trained reviewer

SECONDARY OUTCOMES:
Freezing of Gait Ratio | This outcome will be assessed during in-place turning with and without laser shoes (both collected within the same data collection). The time frame will be 2 hours with or without the lasers followed by 2 hours without or with the lasers.
  Freezing of gait (FoG) ratio is calculated from acceleration of the shins (measured via inertial sensors, Opals by APDM) in-place turning. First, power spectral density from antero-posterior acceleration signals are calculated. Then, a FoG ratio is calculated as the ratio of total power in the "freezing band" (3-8 Hz) and the "locomotion band" (0.5-3 Hz). Higher freezing ratios indicate higher severity of FoG. (Tang et al., 2019).

OTHER OUTCOMES:
Step length during gait | 4 hours
  The step length during gait as quantified by gait map recording.
Foot angle during gait | 4 hours
  The foot angle during gait as quantified by gait map recording.
Foot height during gait | 4 hours
  The foot height during gait as quantified by gait map recording.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy C Ivy, OTD, Principal Investigator — Northern Arizona University
Locations (1):
- Phoenix Biomedical Campus, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tang L, Xu W, Li Z, Chen Y, Chen H, Yu R, Zhu X, Gu D. Quantitative gait analysis for laser cue in Parkinson's disease patients with freezing of gait. Ann Transl Med. 2019 Jul;7(14):324. doi: 10.21037/atm.2019.05.87. PMID 31475194
- [Background] Sejdic E, Fu Y, Pak A, Fairley JA, Chau T. The effects of rhythmic sensory cues on the temporal dynamics of human gait. PLoS One. 2012;7(8):e43104. doi: 10.1371/journal.pone.0043104. Epub 2012 Aug 21. PMID 22927946
- [Result] Barthel C, Nonnekes J, van Helvert M, Haan R, Janssen A, Delval A, Weerdesteyn V, Debu B, van Wezel R, Bloem BR, Ferraye MU. The laser shoes: A new ambulatory device to alleviate freezing of gait in Parkinson disease. Neurology. 2018 Jan 9;90(2):e164-e171. doi: 10.1212/WNL.0000000000004795. Epub 2017 Dec 20. PMID 29263221
- [Result] Ferraye MU, Fraix V, Pollak P, Bloem BR, Debu B. The laser-shoe: A new form of continuous ambulatory cueing for patients with Parkinson's disease. Parkinsonism Relat Disord. 2016 Aug;29:127-8. doi: 10.1016/j.parkreldis.2016.05.004. Epub 2016 May 6. No abstract available. PMID 27161825